CLINICAL TRIAL: NCT02364622
Title: The Effects of Flexible Trachway(R) Intubating Stylet in the Accurate Placement of Left-sided Double-lumen Endobronchial Tube
Brief Title: The Effects of Flexible Intubating Stylet in the Accurate Placement of Double-lumen Endobronchial Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUH-IRB-20130194
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2013-10

CONDITIONS: Intubation Complication; Intubation, Difficult
Keywords: flexible intubating stylet; double-lumen endobronchial tube

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tranditional fiberoptic bronchoscopy (Sham Comparator): The accurate placement of left-sided double lumen endobronchial tube into the left main bronchus was facilitated by traditional fiberoptic bronchoscopy.
  Interventions: Device: Tranditional fiberoptic bronchoscopy
- Modified fiberoptic bronchoscopy (Experimental): The accurate placement of left-sided double lumen endobronchial tube into the left main bronchus was facilitated by modified fiberoptic bronchoscopy.
  Interventions: Device: Modified fiberoptic bronchoscopy
- Flexible Trachway intubating stylet (Experimental): We used Flexible Trachway intubating stylet to facilitate the accurate placement of left-sided double lumen endobronchial tube into the left main bronchus.
  Interventions: Device: Flexible Trachway intubating stylet

INTERVENTIONS:
Device: Tranditional fiberoptic bronchoscopy — The accurate placement of left-sided DLT into the left main bronchus was facilitated by tranditional fiberoptic bronchoscopy.
  Arms: Tranditional fiberoptic bronchoscopy
Device: Modified fiberoptic bronchoscopy — The accurate placement of left-sided DLT into the left main bronchus was facilitated by modified fiberoptic bronchoscopy
  Arms: Modified fiberoptic bronchoscopy
Device: Flexible Trachway intubating stylet — The accurate placement of left-sided DLT into the left main bronchus was faciliated by using flexible Trachway intubating stylet.
  Arms: Flexible Trachway intubating stylet

SUMMARY:
The purpose of this study is to determine whether using the flexible Trachway(R) intubating stylet could facilitate and promote the accurate placement of double-lumen endobronchial tube.

DETAILED DESCRIPTION:
How to accurately place the left-sided double-lumen endobronchial tube (DLT) in the trachea remains a great challenge for anesthesiologists. Although new upper airway devices, such as flexible Trachway (R), a video-assisted intubating stylet, had been developed for facilitating airway management, the larger size and the complexity of DLT makes the difficulties for accurate placement of DLT blindly. Therefore, the investigators designed this study to investigate the effects of flexibleTrachway(R) intubating stylet in the placement of left-sided DLT in the trachea.

ELIGIBILITY:
Inclusion Criteria:

* patients with American Society of Anesthesiologists physical status I-III
* More than 18 years of age
* Requiring DLT for thoracic surgery

Exclusion Criteria:

* risk of regurgitation and pulmonary aspiration
* history of gastroesophageal reflux, pregnancy
* scheduled tracheostomy and postoperative prolonged ventilation in ICU
* patients with limited neck extension (< 35°)
* a distance between the tip of the patient's mandible and hyoid bone of less than 7 cm
* a sternomental distance of less than 12.5 cm with the head fully extended
* mouth can not open

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Main outcome measure is the successful rate of the first accurate placement of left-sided DLT in the trachea | 12 month

SECONDARY OUTCOMES:
The outcome measure is the time needed to accurate placement of left-sided DLT in the trachea | 12 month
The outcome measure is mean blood pressure (MAP) during intubation period | 12 month
  MAP was measured before intubation, and after intubation 1, 3,and 5 min.
The outcome measure is the heart rate (HR) during intubation period | 12 month
  HR was measured and recorded before intubation, and after intubation 1, 3,and 5 min
The outcome measure is the incidence of hypoxemia | 12 month
  Hypoxemia was defined as SPO2 less than 90%. Hypoxemia was recorded during the intubation period.
The outcome measure is the incidence of sore throat | 12 month
  Sore throat was observed and evaluated after extubation and patient regained consciousness
The outcome measure is the incidence of hoarseness | 12 month
  Hoarseness was observed and evaluated after extubation and patient regained consciousness

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Te Hsu, MD, Principal Investigator — Department of Anesthesia, Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Kaohsiung Medical University chung-Ho Memorial Hospital, Kaohsiung City, Taiwan, Taiwan

REFERENCES:
- [Derived] Hsu HT, Kuo YW, Ma CW, Su MP, Tseng KY, Li CL, Cheng KI. Trachway(R) flexible stylet facilitates the correct placement of double-lumen endobronchial tube: a prospective, randomized study. BMC Anesthesiol. 2022 Aug 15;22(1):260. doi: 10.1186/s12871-022-01800-8. PMID 35971080